CLINICAL TRIAL: NCT07225088
Title: DESCANSO/REST (Depresión/Depressed Mood, Cansancio/Fatigue, and Sueño/Sleep): A Trial Assessing Feasibility and Acceptability of an Intervention for Depressed Mood, Insomnia, and Fatigue Symptoms in Latino Cancer Patients
Brief Title: DESCANSO, a Mental Health Intervention for Depression, Insomnia, and Fatigue Symptoms in Latino People With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-277
Record Dates: First submitted 2025-10-15; First posted 2025-11-05 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor; Solid Tumor, Adult
Keywords: Solid Tumor; Solid Tumor Stage I; Solid Tumor Stage II; Solid Tumor Stage III; Memorial Sloan Kettering Cancer Center; 25-277
MeSH Terms: interventions — RE1-silencing transcription factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Intervention: DESCANSO (Experimental): Participants will receive DESCANSO (Depresión/Depressed Mood, Cansancio/Fatigue, and Sueño/Sleep; Rest in English)
  Interventions: Behavioral: DESCANSO/Depresión/Depressed Mood, Cansancio/Fatigue, and Sueño/Sleep; Rest in English
- Control Intervention: Enhanced Usual Care (No Intervention): Participants will receive Enhanced Usual Care

INTERVENTIONS:
Behavioral: DESCANSO/Depresión/Depressed Mood, Cansancio/Fatigue, and Sueño/Sleep; Rest in English — DESCANSO (Depresión/Depressed Mood, Cansancio/Fatigue, and Sueño/Sleep; Rest in English)
  Arms: Experimental Intervention: DESCANSO

SUMMARY:
The purpose of this study is to improve ways of providing mental health support to Spanish-speaking Latino participants who have cancer and experience depression, insomnia, and fatigue. Investigators will test a special mental health intervention called DESCANSO/REST (Depresión/Depressed Mood, Cansancio/Fatigue, and Sueño/Sleep). The intervention can be delivered through telehealth.

ELIGIBILITY:
Provider Eligibility Criteria:

Participant eligibility will be determined by a self-report screener. Inclusion Criteria Self-Report Criteria

* Mental health provider
* Treats Latino cancer patients and/or survivors
* Has at least 3 years of clinical experience providing psychosocial services to cancer patients and/or survivors
* Able to read Spanish determined by the question: "Can you read in Spanish? Yes/No"

Patient Eligibility Criteria:

A patient cannot be considered eligible for this study unless ALL of the following conditions are met. Participant eligibility will be determined by an initial EMR review followed by a self-report screener.

Inclusion Criteria EMR Criteria

* Documentation of Disease

  o Pathologically confirmed solid tumor cancer (either most recent or new diagnosis)
* Definition of Disease [or Measurable Disease]

  o Diagnosed with stages I, II, or III
* Prior Treatment

  * Currently undergoing systemic therapy (chemotherapy, radiation therapy, and/or immunotherapy) or within the first year following completion of systemic therapy Self-Report Criteria
  * Age ≥ 21 years
  * Lives in mainland U.S. or Puerto Rico
  * Identifies as Latino/a or Hispanic
  * Reports Spanish as their preferred language
  * Speaks Spanish "Very well" or "Well" as determined by the question: "How well do you speak Spanish?"
  * Presence of fatigue and disturbed sleep determined by a score of ≥ 3 on the MD Anderson Symptom Inventory

Exclusion Criteria EMR Criteria

o In the judgment of the treating physician, protocol investigators, and/or study staff, presence of cognitive impairment (e.g., delirium or dementia) sufficient to preclude meaningful informed consent and/or study participation

Self-Report Criteria

* History of comorbidities within the last 12 months associated with fatigue and poor sleep, including hypothyroidism or abnormal thyroid function, sleep apnea, chronic obstructive pulmonary disease, neuromuscular disease, alcohol or drug abuse
* Pregnant or lactating, women only
* Presence of suicidal risk determined by any affirmative response on the Columbia-Suicide Severity Rating Scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2026-01-23 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants who complete at least 5 DESCANSO sessions | Up to 1 year
  Feasibility of DESCANSO (Depresión/Depressed Mood, Cansancio/Fatigue, and Sueño/Sleep) defined as completing at least 5 out of the planned 8 DESCANSO sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Rosario Costas Muniz, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Cancer Center Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited protocol activity), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
• Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org